CLINICAL TRIAL: NCT01536444
Title: Use of the Epidermal Expansion System to Harvest and Place Suction Blister Epidermal Grafts on Wounds in Patients After Mohs or Excisional Surgery for Skin Cancer
Brief Title: Use of the Epidermal Micrografts for Wound Healing After Mohs or Excisional Surgery for Skin Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Momelan Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-DMG-1
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Neoplasm of Skin
Keywords: Mohs surgery; Excisional skin surgery; Micrografting
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micrografting (Experimental)
  Interventions: Device: Momelan Technologies Epidermal Graft Harvesting System

INTERVENTIONS:
Device: Momelan Technologies Epidermal Graft Harvesting System — The procurement of the epidermal micrograft involves the use of the MoMelan Technologies suction blister system which consists of a control box that creates the vacuum necessary to create the microblisters and a harvester. The device is applied to the subject's thigh to create blisters. The epidermal micrografts are then harvested and transferred to Tegaderm™ and then placed on the surgical wound and the wound is bandaged.

SUMMARY:
This case series will assess the use of suction blister epidermal grafts harvested by a novel device on select patients that have wounds from Mohs or excisional surgery.

DETAILED DESCRIPTION:
This study evaluates a novel micrografting technique to determine how it will influence the healing and cosmetic result of selected post surgical wounds in 12 subjects. The Epidermal Expansion System (designed by MoMelan Technologies) will generate an array of small microblisters and transfer the micrografts to a sterile wound dressing for application to the subject's surgical area. The sponsor hypothesizes that applying expanded micrografts to wounds that otherwise would have healed by second intention alone will hasten healing and possibly reduce scarring.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females between 35 and 90 years of age
* Status post skin cancer removal on the scalp, ear or leg with a wound that would otherwise be allowed to heal by secondary intention or grafting
* Wound considered appropriate by physician to receive epidermal grafting
* Willingness to participate in study by evidence of informed consent

Exclusion Criteria:

* Female patients reported to be breastfeeding, pregnant or planning to become pregnant
* Clinical signs of infection
* Subjects currently on immunosuppressive medications, chemotherapy or a cytotoxic agent
* Participation in another interventional study with potential exposure to an investigational drug or device within the past 30 days or planned study entry within 90 days after study entrance.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Wound healing/scarring | 6 weeks

SECONDARY OUTCOMES:
Incidence of adverse events | 6 weeks
Physician global satisfaction | 6 weeks
Subject global satisfaction | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashish C. Bhatia, MD, Principal Investigator — DuPage Medical Group
Locations (1):
- DuPage Medical Group, Naperville, Illinois, United States